CLINICAL TRIAL: NCT06436157
Title: Genetic Testing Uptake Through an Enhanced Oncology Nurse-Led Intervention in Patients With Solid Tumors (GENESIS): A Pilot Study
Brief Title: A Pilot Study of Genetic Testing Uptake Through Enhanced Oncology Nurse-Led Intervention
Acronym: GENESIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Enloe Regional Cancer Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GENESIS
Record Dates: First submitted 2024-05-15; First posted 2024-05-30 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumor, Adult
Keywords: Genetic Counseling and Testing; NCCN guidelines; Utilization; Feasibility; Nurse-led care coordination
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: This pilot study will randomize patients who are starting or switching their systemic therapies for solid cancers, eligible for GCT, and have not undergone prior genetic testing into two groups: "enhanced education intervention" and "usual care education".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Education Intervention (Experimental): Patients in the enhanced education intervention arm will be scheduled for a redesigned therapy education session with a trained oncology nurse.
  Interventions: Other: Enhanced education
- Usual Care Education Arm (Active Comparator): Patients in this arm will receive the usual care education provided to cancer patients undergoing systemic therapy, which includes information on treatment options, side effects, and support services without targeted genetic testing education.
  Interventions: Other: Usual care education

INTERVENTIONS:
Other: Enhanced education — In addition to the education conducted as part of usual care, the nurse will: 1) provide basic education on GCT; and 2) if the patient is eligible and agreeable to GCT, place a referral to GCT (if not already ordered).
  Patients will also be provided with written materials reinforcing the key messages of GCT education, designed to be understandable to individuals without a medical background. Nurses will also conduct a follow-up "nudge" by sending an in basket message via electronic medical record to ensure that the referrals are processed by the referral coordinators.
  Arms: Enhanced Education Intervention
Other: Usual care education — A brief introduction to GCT will be provided in accordance with the information covered in the "chemo education binder," which is the current standard of care at Enloe Regional Cancer Center. As per the usual care, referrals for genetic testing will be clinician-initiated without the proactive involvement of the RN.
  Arms: Usual Care Education Arm

SUMMARY:
Genetic factors are a significant determinant of the likelihood of developing various types of cancers. Identification of germline risk can have important implications for both patients and their families. Although estimates vary, pathogenic germline variants can be seen in ~3-17.5% of unselected patients with cancer with important clinical significance. Unfortunately, despite progress in multigene testing and the identification of heritable conditions, genetic counseling and testing (GCT) remains underutilized among cancer patients. Although there are multiple barriers to low testing, initial referral to GCT from the treating oncologist has been noted to be the most significant barrier.

Nurse navigation has been shown to improve the timeliness of cancer care and patient outcomes across various cancer types and improve the uptake of genomic testing in cancer patients. Despite proven benefits, community cancer centers often face resource limitations that prevent them from consistently assigning a dedicated nurse navigator to cancer patients. However, community centers universally have oncology nurses who routinely educate patients about their systemic therapies. By enhancing the "therapy education" sessions, the investigators hypothesize that oncology nurses can bridge this gap and potentially identify eligible patients, provide essential education on the importance of genetic testing, and facilitate the referral process. The investigators propose a pilot randomized study to evaluate the potential effectiveness, acceptability, and feasibility of a novel, nurse-led "enhanced education" intervention specifically designed to increase the uptake of GCT in adult cancer patients.

DETAILED DESCRIPTION:
Identification of germline risk can have important implications for both patients and their families: it can help patients develop tailored cancer surveillance, risk-reducing measures, reproductive planning, identify novel genotype-directed drug targets, and also optimally address the risk of malignancy in at-risk relatives. Although estimates vary, pathogenic germline variants (PGV) can be seen in ~3-17.5% of unselected patients with cancer with important clinical significance. Although national and international guidelines such as the National Comprehensive Cancer Network (NCCN) outline the criteria for who should be offered genetic counseling and testing (GCT) based on a patient's personal and/or family history, recent studies have found that broader testing of at-risk patients might help identify PGV in patients who otherwise would not have met guidelines for genetic testing.

Unfortunately, despite progress in multigene testing and the identification of heritable conditions, GCT remains underutilized among cancer patients. A recent study revealed that the uptake of germline testing among cancer patients remains strikingly low; in California and Georgia, between 2013 and 2019, less than 7% of patients diagnosed with cancer underwent such testing. While a study indicates a promising recent increase in the use of germline testing among women diagnosed with breast and ovarian cancer from 2012 to 2019, there is still a significant gap in ensuring that all eligible patients are provided with GCT. Although there are multiple barriers to low testing, initial referral to GCT from the treating oncologist has been noted to be the most significant barrier.

Community cancer centers are crucial in providing accessible care to a large segment of the cancer patient population. However, community cancer centers often face various challenges with limited resources for specialized genetic services variability in community oncologists' practice patterns and perceptions in GCT, and potentially urban-rural variability in patient awareness and understanding of the potential impact of genetic testing on their care.

Nurse navigation has been shown to improve the timeliness of cancer care and patient outcomes across various cancer types, in addition to improving the uptake of genomic testing in cancer patients. Despite proven benefits, community cancer centers often face resource limitations that prevent them from consistently assigning a dedicated nurse navigator to cancer patients. However, community centers universally have oncology nurses who routinely educate patients about their systemic therapies. By enhancing the "therapy education" sessions, the investigators hypothesize that oncology nurses can bridge this gap and potentially identify eligible patients, provide essential education on the importance of genetic testing, and facilitate the referral process. This approach leverages the trust and communication between nurses and patients and the principle that informed patients are more likely to engage in their healthcare decisions to potentially overcome barriers to genetic testing uptake.

The investigators propose a pilot randomized study to evaluate the potential effectiveness, acceptability, and feasibility of a novel, nurse-led "enhanced education" intervention specifically designed to increase the uptake of GCT in adult cancer patients. Patients in the enhanced education arm will be scheduled for an enhanced therapy education session with a trained oncology nurse for patients starting or switching their systemic therapies. In addition to the education conducted as part of the usual care, the nurse will: 1) provide detailed education on GCT; and 2) if the patient is eligible and agreeable to GCT, order a referral to GCT (if not already ordered). Nurses will provide a "nudge" to the referral coordinators within a week of the education session to ensure the referral process is completed.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years)
* Diagnosed with a solid tumor cancer type that has established guidelines suggesting the utility of genetic testing in treatment (breast, ovarian, prostate, pancreatic, colon, Lynch syndrome-related cancers (colorectal, endometrial, gastric, ovarian, pancreatic, urothelial, brain (usually glioblastoma), biliary tract, small intestine), Li-Fraumeni syndrome tumor spectrum (e.g., soft tissue sarcoma, osteosarcoma, central nervous system tumors, breast cancer, adrenocortical carcinoma), etc.)
* Eligible for GCT based on the current NCCN guidelines
* Starting new systemic therapy or switching systemic therapy
* Eligible for GCT as per the current NCCN guidelines
* No prior genetic testing (or tested before 2014)

Exclusion Criteria:

* Prior GCT with test results available (if tested 2014 onwards)
* Patients scheduled for treatment education with Advanced Practice Provider (typically reserved for more complex regimens)
* Patients with cognitive impairments or severe psychological disorders that would limit their ability to understand the genetic counseling/testing information or give informed consent.
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures (e.g., patients requiring urgent therapy and/or inpatient chemotherapy initiation).
* Patients who are currently participating in other clinical trials that could confound the outcomes of genetic testing uptake.
* Prospective participants who, in the investigator's opinion, may not be able to comply with all study procedures (including compliance issues related to logistics).
* Hematologic malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2025-03-26 (Estimated); Study Completion 2025-09-26 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients in each arm who proceed to GCT consultation following the intervention. | Through study completion, an average of 9 months

SECONDARY OUTCOMES:
Percentage of patients in each arm referred to GCT | Through study completion, an average of 9 months
Average time from GCT referral order to GCT consultation | Through study completion, an average of 9 months
Average time from GCT consultation to completion of genetic testing | Through study completion, an average of 9 months

OTHER OUTCOMES:
Recruitment rates, completion rate of follow-up assessments, and retention rates. | Through study completion, an average of 9 months
  Recruitment rates (percentage of participants who agree to participate out of those approached), completion rate of follow-up assessments (percentage of patients that complete follow-up assessment), and retention rates (percentage of patients retained in the study throughout the study period).
Average scores on the AIM post intervention | Within 3 weeks of nursing education intervention
Average scores and qualitative feedback from post-intervention survey questionnaire to measure satisfaction with the study and recommendations for improvement from participants, nurses and genetic counselors | Within 3 weeks of nursing education intervention and through study completion, an average of 9 months
RN workload as measured by average time spent per patient and perception (Likert-scale-based and qualitative feedback) | Through study completion, an average of 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Ranjan Pathak, MD MHS, Principal Investigator — Enloe Health
Locations (2):
- United States (2):
  - Enloe Regional Cancer Center, Chico, California
  - University of California, Davis, Sacramento, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurian AW, Abrahamse P, Furgal A, Ward KC, Hamilton AS, Hodan R, Tocco R, Liu L, Berek JS, Hoang L, Yussuf A, Susswein L, Esplin ED, Slavin TP, Gomez SL, Hofer TP, Katz SJ. Germline Genetic Testing After Cancer Diagnosis. JAMA. 2023 Jul 3;330(1):43-51. doi: 10.1001/jama.2023.9526. PMID 37276540
- [Background] Daly MB, Pal T, Maxwell KN, Churpek J, Kohlmann W, AlHilli Z, Arun B, Buys SS, Cheng H, Domchek SM, Friedman S, Giri V, Goggins M, Hagemann A, Hendrix A, Hutton ML, Karlan BY, Kassem N, Khan S, Khoury K, Kurian AW, Laronga C, Mak JS, Mansour J, McDonnell K, Menendez CS, Merajver SD, Norquist BS, Offit K, Rash D, Reiser G, Senter-Jamieson L, Shannon KM, Visvanathan K, Welborn J, Wick MJ, Wood M, Yurgelun MB, Dwyer MA, Darlow SD. NCCN Guidelines(R) Insights: Genetic/Familial High-Risk Assessment: Breast, Ovarian, and Pancreatic, Version 2.2024. J Natl Compr Canc Netw. 2023 Oct;21(10):1000-1010. doi: 10.6004/jnccn.2023.0051. PMID 37856201
- [Background] Kurian AW, Ward KC, Abrahamse P, Bondarenko I, Hamilton AS, Deapen D, Morrow M, Berek JS, Hofer TP, Katz SJ. Time Trends in Receipt of Germline Genetic Testing and Results for Women Diagnosed With Breast Cancer or Ovarian Cancer, 2012-2019. J Clin Oncol. 2021 May 20;39(15):1631-1640. doi: 10.1200/JCO.20.02785. Epub 2021 Feb 9. PMID 33560870
- [Background] Swink A, Nair A, Hoof P, Matthews A, Burden C, Johnson K, Blum JL. Barriers to the utilization of genetic testing and genetic counseling in patients with suspected hereditary breast and ovarian cancers. Proc (Bayl Univ Med Cent). 2019 Jun 11;32(3):340-344. doi: 10.1080/08998280.2019.1612702. eCollection 2019 Jul. PMID 31384183
- [Background] McAllister KA, Schmitt ML. Impact of a nurse navigator on genomic testing and timely treatment decision making in patients with breast cancer. Clin J Oncol Nurs. 2015 Oct;19(5):510-2. doi: 10.1188/15.CJON.510-512. PMID 26414569
- [Background] Rives TA, Pavlik H, Li N, Qasrawi L, Yan D, Pickarski J, Dietrich CS, Miller RW, Ueland FR, Kolesar JM. Implementation of Nurse Navigation Improves Rate of Molecular Tumor Testing for Ovarian Cancer in a Gynecologic Oncology Practice. Cancers (Basel). 2023 Jun 15;15(12):3192. doi: 10.3390/cancers15123192. PMID 37370804
- [Background] DiBiase JF, Scharnetzki E, Edelman E, Lucas FL, Helbig P, Rueter J, Han PKJ, Ziller E, Jacobs EA, Anderson EC; MCGI Working Group. Urban-Rural and Socioeconomic Differences in Patient Knowledge and Perceptions of Genomic Tumor Testing. JCO Precis Oncol. 2023 Mar;7:e2200631. doi: 10.1200/PO.22.00631. PMID 36893376
- [Background] Anderson EC, Hinton AC, Lary CW, Fenton ATHR, Antov A, Edelman E, Helbig P, Reed K, Miesfeldt S, Thomas CA, Hall MJ, Roberts JS, Rueter J, Han PKJ; MCGI Working Group. Community oncologists' perceptions and utilization of large-panel genomic tumor testing. BMC Cancer. 2021 Nov 25;21(1):1273. doi: 10.1186/s12885-021-08985-0. PMID 34823486
- [Background] Idos GE, Kurian AW, Ricker C, Sturgeon D, Culver JO, Kingham KE, Koff R, Chun NM, Rowe-Teeter C, Lebensohn AP, Levonian P, Lowstuter K, Partynski K, Hong C, Mills MA, Petrovchich I, Ma CS, Hartman AR, Allen B, Wenstrup RJ, Lancaster JM, Brown K, Kidd J, Evans B, Mukherjee B, McDonnell KJ, Ladabaum U, Ford JM, Gruber SB. Multicenter Prospective Cohort Study of the Diagnostic Yield and Patient Experience of Multiplex Gene Panel Testing For Hereditary Cancer Risk. JCO Precis Oncol. 2019 Mar 28;3:PO.18.00217. doi: 10.1200/PO.18.00217. eCollection 2019 Mar. PMID 34322651
- [Background] Samadder NJ, Riegert-Johnson D, Boardman L, Rhodes D, Wick M, Okuno S, Kunze KL, Golafshar M, Uson PLS Jr, Mountjoy L, Ertz-Archambault N, Patel N, Rodriguez EA, Lizaola-Mayo B, Lehrer M, Thorpe CS, Yu NY, Esplin ED, Nussbaum RL, Sharp RR, Azevedo C, Klint M, Hager M, Macklin-Mantia S, Bryce AH, Bekaii-Saab TS, Sekulic A, Stewart AK. Comparison of Universal Genetic Testing vs Guideline-Directed Targeted Testing for Patients With Hereditary Cancer Syndrome. JAMA Oncol. 2021 Feb 1;7(2):230-237. doi: 10.1001/jamaoncol.2020.6252. PMID 33126242
- [Background] Teresi JA, Yu X, Stewart AL, Hays RD. Guidelines for Designing and Evaluating Feasibility Pilot Studies. Med Care. 2022 Jan 1;60(1):95-103. doi: 10.1097/MLR.0000000000001664. PMID 34812790